CLINICAL TRIAL: NCT05123417
Title: Comparison of Nursing Students' Knowledge Levels on Pressure Ulcer Prevention Using Flipped Learning and Traditional Learning Models: A Randomized Controlled Study
Brief Title: Knowledge and Practices of Preventing Pressure Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Kerem Yıldız, Principal Investigator, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ETK00-2022-0021
Record Dates: First submitted 2021-10-15; First posted 2021-11-17 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Pressure Ulcer
Keywords: Pressure Ulcer Prevention; Kowledge; Nursing Student
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Single (Care Provider)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention group students will be educated with educational materials (lecture presentation, video) will be uploaded through the system in accordance with the flipped learning model, and students will be asked to come prepared to the planned lesson. No classical presentations will be made to the students, but the education will be carried out in the form of question and answer discussion, in line with the Flipped Learning model. After the lesson, the questions of the students who have questions will be answered.
  Interventions: Diagnostic Test: Follow up
- Control Group (No Intervention): The training, consisting of control group students will be trained with Powerpoint presentation, which will last 20-30 on average, will be given in accordance with the traditional education model. After the lesson, the questions of the students who have questions will be answered.

INTERVENTIONS:
Diagnostic Test: Follow up — Each group participants will be tested with questionnaire before the training and two weeks after the training they will get post test with the same questionnaire.
  Arms: Intervention Group

SUMMARY:
Pressure ulcer is defined by the European Pressure Ulcer Advisory Panel (EPUAP) and the National Pressure Ulcer Advisory Panel (NPUAP) as "localized skin and/or skin, usually arising over bony prominences, caused by pressure alone, or by a combination of shear and pressure. subcutaneous tissue damage. Pressure ulcer is a painful, costly and preventable health problem that is frequently encountered especially in geriatrics group and in patients with limited daily activities or bedridden. It is an undesirable health care problem that is difficult to treat, but it is possible to prevent the development of pressure ulcers with the measures to be taken from the beginning of the disease. In order for nurses to fulfill their role in preventing pressure ulcers, the content of undergraduate education programs needs to be arranged in a way that will provide them with knowledge and skills in the prevention of pressure ulcers, diagnosis of risky patients and maintenance of care. In Northern Cyprus, knowledge and skills related to pressure sores are provided to students in the basic nursing education curriculum. However, the subject of pressure ulcer in the education programs of nursing schools differs in terms of content and duration, and most of the hospitals do not have a standard guide and training program for the prevention of pressure ulcers. In Northern Cyprus, studies on the knowledge and practices of nursing students to prevent pressure ulcers are limited. According to the results of a study conducted in Turkey, it has been reported that a significant portion of nursing students have a positive attitude towards preventing pressure ulcers, but their general knowledge about preventing pressure ulcers is insufficient. In another study, it was reported that 70.7% of nursing students encountered patients with pressure ulcers during hospital practices, but research findings and the knowledge of nursing students to prevent the development of pressure ulcers were insufficient. Similarly, in studies conducted with nursing students using different scales, it has been reported that students' knowledge levels about preventing pressure ulcers are low. This research was planned in accordance with the randomized controlled research method in order to determine the knowledge levels and practices of firts year nursing students to prevent pressure ulcers.

DETAILED DESCRIPTION:
The population of the research will be 2nd year students studying at the Faculty of Health Sciences Nursing Department in the 2021-2022 Academic Year Spring Semester. Since 1st year students do not have any information about pressure ulcers yet and other classes (3rd, 4th grade students) have received information about pressure ulcers before, they were excluded from the study, as this would affect the average scores. The entire population that meets the criteria for inclusion in the study will be included in the sample. Before starting the research, the enclosed Informed Consent Form will be distributed to the students and their consent will be obtained stating that they are willing to participate in the research. "Student Descriptive Characteristics Questionnaire and "Pressure ulcer Knowledge Assessment Tool" updated version (PUKAT 2.0) all groups will be collected before and after the training by face-to-face interview method. Students will be divided into two groups by simple randomization method. Group distributions will be divided into group 1 and group 2 by drawing lots. Students who are divided into groups will not know what the group they belong to means In this case, group 1 students will be included in the research in accordance with the flipped learning model, and group 2 students will be included in the research in accordance with the traditional education method. Group 1 students and educational materials (lecture presentation, video) will be uploaded through the system in accordance with the flipped learning model, and students will be asked to come prepared to the planned lesson. No classical presentations will be made to the students, but the education will be carried out in the form of question and answer discussion, in line with the Flipped Learning model. The training, consisting of Group 2 students and a Powerpoint presentation, will last 20-30 on average, and will be given in accordance with the traditional education model. After the lesson, the questions of the students who have questions will be answered. After obtaining the necessary ethics committee approval, the data collection phase will begin.

ELIGIBILITY:
Inclusion Criteria:

* Students who agree to participate in the research,
* Year 2 students studying at the University's Faculty of Health Sciences, Department of Nursing.

Exclusion Criteria:

* Students who do not meet the sample selection criteria,
* Students who fill in the data collection form incompletely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Knowledge Evaluation Scale for Pressure Ulcer Prevention From | 2 weeks
  Students will fill the Knowledge Evaluation Scale for Pressure Ulcer Prevention From during the pre-test phase. Then, post-test was applied 2 weeks after the necessary training models were applied. Students will ve evaluate with minimum 0 points, maximum 25 points over Knowledge Evaluation Scale for Pressure Ulcer Prevention From.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dag Sucu G, Firat Kilic H. Knowledge and attitudes of Turkish nursing students towards pressure injury prevention. J Tissue Viability. 2022 Feb;31(1):16-23. doi: 10.1016/j.jtv.2021.08.003. Epub 2021 Aug 25. PMID 34462179
- [Result] Edsberg LE, Black JM, Goldberg M, McNichol L, Moore L, Sieggreen M. Revised National Pressure Ulcer Advisory Panel Pressure Injury Staging System: Revised Pressure Injury Staging System. J Wound Ostomy Continence Nurs. 2016 Nov/Dec;43(6):585-597. doi: 10.1097/WON.0000000000000281. PMID 27749790
- [Result] Reddy M, Gill SS, Rochon PA. Preventing pressure ulcers: a systematic review. JAMA. 2006 Aug 23;296(8):974-84. doi: 10.1001/jama.296.8.974. PMID 16926357
- [Result] Akyol AD. Intervention studies for prevention of pressure ulcers in Turkey: a literature review. Int Nurs Rev. 2006 Dec;53(4):308-16. doi: 10.1111/j.1466-7657.2006.00503.x. PMID 17083421
- [Result] Kisacik OG, Sonmez M. Pressure ulcers prevention: Turkish nursing students' knowledge and attitudes and influencing factors. J Tissue Viability. 2020 Feb;29(1):24-31. doi: 10.1016/j.jtv.2019.11.003. Epub 2019 Nov 10. No abstract available. PMID 31759832
- [Result] Yilmazer T, Tuzer H, Inkaya B, Elcin M. The impact of standardized patient interactions on nursing students' preventive interventions for pressure ulcers. J Tissue Viability. 2020 Feb;29(1):19-23. doi: 10.1016/j.jtv.2019.11.004. Epub 2019 Nov 15. PMID 31757581
- [Result] Dalli OE, Yildirim Y, Caliskan G, Girgin NK. Reliability and validity of the Turkish version of pressure ulcer knowledge assessment tool-updated version (PUKAT 2.0). J Tissue Viability. 2022 Feb;31(1):52-57. doi: 10.1016/j.jtv.2021.08.001. Epub 2021 Aug 11. PMID 34429220